CLINICAL TRIAL: NCT04262739
Title: Open-label, Phase I Clinical Trial to Assess the Maximum Tolerated Dose (MTD), Safety and Efficacy of NYH817G and NYH100P in Monotherapy and Combination in Patients With Advanced Solid Tumors Who Have Failed Approved Standard Therapies
Brief Title: MTD, Safety and Efficacy of NYH817G and NYH100P in Monotherapy and Combination in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haim Bio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HBCR-GP-01
Record Dates: First submitted 2020-02-02; First posted 2020-02-10 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-04

CONDITIONS: Advanced Solid Tumors
Keywords: solid tumors; failed approved standard therapies; advanced solid tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NYH817G (Experimental)
  Interventions: Drug: NYH817G
- NYH100P (Experimental)
  Interventions: Drug: NYH100P
- NYH817G and NYH100P (Experimental)
  Interventions: Drug: NYH817G and NYH100P

INTERVENTIONS:
Drug: NYH817G — Subject will orally administer NYH817G (15 mg) during the cycles(21 days)
  Arms: NYH817G
Drug: NYH100P — Subject will orally administer NYH100P (100 mg) during the cycles(21 days)
  Arms: NYH100P
Drug: NYH817G and NYH100P — Subject will orally administer NYH817G (15 mg) and NYH100P (100 mg) during the cycles(21 days)
  Arms: NYH817G and NYH100P

SUMMARY:
The objectives of this study are:

Part 1:

* To assess the MTD, safety and efficacy of each NYH817G and NYH100P in monotherapy in patients with advanced solid tumors who have failed approved standard therapies.
* To assess the PK properties and the preliminary effectiveness of monotherapy of NYH817G and NYH100P.

Part 2:

* To assess the MTD, RP2D, safety and efficacy of NYH817G and NYH100P in combination therapy in patients with advanced solid tumors who have failed approved standard therapies
* To assess the PK properties, the preliminary effectiveness and the changes in metabolism of combination therapy of NYH817G and NYH100P.

ELIGIBILITY:
Inclusion Criteria:

* 19+ years old
* Diagnosed with advanced solid tumor histologically/cytologically
* Patient without standard therapies or who have failed approved standard therapies
* Those with a disease that is measurable and/or evaluable with the appropriate imaging examination according to RECIST v1.1
* ECOG performance status 0 to 2
* Patients with the suitable marrow, kidney, liver functions, blood coagulation and glycemic control functions
* Patients whose Life expectancy is over 12 weeks
* Patients who signed the agreement to voluntarily participate in this study

Exclusion Criteria:

* Patients who have received a major surgery, radiotherapy, chemotherapy, biologic therapy, targeted therapy, cancer immunotherapy or metabolic therapy within specified weeks counting from the initial administration of the IPs
* Diagnosed with a malignant tumor other than the relevant disease in the last 5 years from the initial administration of the IPs
* Toxicity level has not been recovered to CTCAE Grade 1 or lower
* Has uncontrolled metastasis to the CNS
* Suspected of having a serious infectious disease, paralysis of intestine, bowel obstruction, interstitial pneumonia or pulmonary fibrosis
* Had serious GI bleed or a disease that may affect the absorption of the oral drug in the past 4 weeks
* Considered as having a serious heart disease by the investigator or a serious internal disease
* Has administered a drug from another study within 4 weeks
* Has administered live vaccines within 4 weeks
* Has abused substance or alcohol within 12 weeks
* Has a serious trauma
* Has a history or currently has a type 1 or 2 diabetes
* Has a history of lactic acidosis
* Has glucose-6-phosphate dehydrogenase deficiency
* Has HIV or active or an active hepatitis B or C
* Has a history of psychological condition that could threaten observation of this protocol
* Has a history of hypersensitive reaction to the main ingredient or component of the IP or biguanide class drugs
* Being pregnant or a lactating woman, or (+) pregnancy test
* A female subject of a childbearing age who plans to get pregnant or disagrees to use recommended contraceptions
* Has not agreed to abstain from alcohol
* Considered as unsuitable for the study for other reason by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Safety assessment: Adverse event | Up to 2 years
  Number of adverse events as assessed by NCI CTCAE v5.0
Effectiveness assessment: Disease control rate | Up to 2 years
  To assess the clinical efficacy associated wtih the administration of NYH817G and NYH100P according to the RECIST v1.1

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Parameter: Cmax of NYH817G and NYH100P | At the start and end of Cycle 1 (each cycle is 21 days)
  Cmax is defined as the maximum observed concentration of each drug

OTHER OUTCOMES:
Metabolite change-related: ALDH (for Part 2) | At the start and end of Cycle 1 (each cycle is 21 days)
  To evaluate activity of metabolism in tumor tissues
Metabolism imaging marker-related (for Part 2) | At the start and end of Cycle 1 (each cycle is 21 days)
  FDG PET-CT (Fluorodeoxyglucose Positron Emission Tomography-Computed Tomography)

CONTACTS AND LOCATIONS:
Overall Officials: Minkyu Jung., MD.,Ph.D., Principal Investigator — Div. of Medical Oncology. Yonsei Cancer Center.
Locations (1):
- Severance Hospital, Seoul, South Korea